CLINICAL TRIAL: NCT03267199
Title: The Relationship Between Mean Platelet Volume , Platelet Distribution Width , Platelet Function and ST Segment Resolution in STEMI Patients Treated With Either Thrombolytic Therapy or Primary Percutaneous Coronary Intervention
Brief Title: The Relationship Between MPV,PDW,PFT and ST Segment Resolution in STEMI Patients Treated With Thrombolytic or Primary PCI
Status: Withdrawn | Type: Observational
Why Stopped: Another study was done instead
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nardeen Beshay, resident physician, Assiut University
Other Study IDs: 17100302
Record Dates: First submitted 2017-08-25; First posted 2017-08-30 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: STEMI - ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Fibrinolytic Agents; Blood Cell Count; Platelet Function Tests; Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with high MPV,PDW,PFT: patients with high MPV,PDW,platelet function test
  Interventions: Drug: Thrombolytic; Procedure: Primary PCI; Diagnostic Test: Complete blood count; Diagnostic Test: Platelet function test; Diagnostic Test: ECG
- patients with normal or low MPV,PDW, PFT: patients with normal or low MPV,PDW,platelet function test
  Interventions: Drug: Thrombolytic; Procedure: Primary PCI; Diagnostic Test: Complete blood count; Diagnostic Test: Platelet function test; Diagnostic Test: ECG

INTERVENTIONS:
Drug: Thrombolytic — Thrombolytic therapy
Procedure: Primary PCI — Primary percutaneous coronary intervention
Diagnostic Test: Complete blood count — Blood sample for complete blood count
Diagnostic Test: Platelet function test — Blood sample for platelet function test
Diagnostic Test: ECG — Electrocardiogram

SUMMARY:
* The relationship between admission MPV, PDW, platelet function test and ST-segment resolution in STEMI patients treated with either thrombolytic therapy or primary percutaneous coronary intervention
* The relationship between admission MPV, PDW, platelet function test and high thrombus burden & post-PCI Thrombolysis In Myocardial Infarction (TIMI) flow of infarct related artery in STEMI patients treated with primary percutaneous coronary intervention

DETAILED DESCRIPTION:
Reperfusion therapy as the main treatment strategy in patients with ST-segment elevation myocardial infarction (STEMI) consists of either thrombolysis or primary percutaneous coronary intervention (pPCI). Primary percutaneous coronary intervention is the preferred therapy for STEMI; however, cardiac catheterization laboratories may not be widely available.

Early recanalization of the infarct related artery (IRA) by either thrombolytics or percutaneous coronary intervention (PCI) is the main goal in the treatment of acute myocardial infarction. But the eventual aim is to provide reperfusion at the tissue level as well as in the infarct related artery .

Resolution of ST elevation has been shown as an agreeable marker that reflects both epicardial and myocardial reperfusion . In addition, early and complete resolution of ST -segment in the setting of acute myocardial infarction is associated with smaller infarct size, greater ejection fraction and reduced morbidity and mortality .

Platelets play a critical role in the pathogenesis and prognosis of ACS . They secrete a number of substances that are key mediators of coagulation, thrombosis and atherosclerosis. High-volume platelets have a higher thrombotic potential than small platelets and have concentrated granule contents that are of interest in the development of ACS pathogenesis . Mean platelet volume (MPV) is the most commonly used measure of platelet size and correlates with platelet activity. Platelet distribution width (PDW) is an index reflecting heterogeneous platelet size, whereas the platelet-large cell ratio (P-LCR) is the proportion of large platelets in blood circulation. Generally, higher MPV, PDW and P-LCR are correlated with increased platelet size, although they tend to be overlooked in clinical applications. In fact, these indices, particularly MPV and PDW, correlate with platelet functions.

Percutaneous coronary intervention (PCI) is an effective treatment for acute coronary syndrome (ACS), including ST-elevation myocardial infarction (STEMI) and unstable angina. Despite the efficacy of the technique, preprocedural high-thrombus burden (HTB) is a predictor of procedural complications following primary PCI for STEMI. HTB can lead to poor outcomes, including distal embolization, no-reflow, increased myocardial necrosis and decreased left ventricular function.

Although MPV is associated with impaired angiographic reperfusion and poor clinical outcome in patients with STEMI,little is known regarding the association between MPV levels and infarct related artery patency in those patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with STEMI presented who will be treated with either thrombolytic therapy or primary PCI in assiut university cath lab will be included in the study

Exclusion Criteria:

* Patient with complete LBBB on admission ECG
* Active infection
* Documented systemic inflammatory disease
* Malignancy
* End-stage liver
* Renal failure
* Patient receiving oral anticoagulation medicine
* Bleeding diathesis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with STEMI presented who will be treated with either thrombolytic therapy or primary PCI in assiut university cath lab will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Correlation between admission MPV ,PDW ,platelet function test and change in ST-segment elevation in STEMI patients assessed by CBC ,platelet function test & ECG | Baseline and 90 min after either the beginning treatment with thrombolytic therapy or primary PCI
  Correlation between admission MPV ,PDW ,platelet function test and change in ST-segment elevation in STEMI patients treated with either thrombolytic therapy or primary percutaneous coronary intervention assessed by CBC,platelet function test & ECG

SECONDARY OUTCOMES:
Correlation between MPV,PDW,platelet function test and TIMI flow of infarct related artery in STEMI patients treated with primary PCI | Baseline
  Correlation between MPV ,PDW,platelet function test and post-PCI Thrombolysis In Myocardial Infarction (TIMI) flow of infarct related artery in STEMI patients treated with primary percutaneous coronary intervention
Correlation between MPV,PDW,platelet function test and high thrombus burden of infarct related artery in STEMI patients treated with primary PCI | Baseline
  Correlation between MPV ,PDW,platelet function test and high thrombus burden of infarct related artery in STEMI patients treated with primary percutaneous coronary intervention